CLINICAL TRIAL: NCT00041561
Title: The Effects of Inhaled Nitric Oxide in the Treatment of Acute Hypoxemic Respiratory Failure (AHRF) In Pediatrics
Brief Title: Effects of Inhaled Nitric Oxide in the Treatment of Acute Hypoxemic Respiratory Failure (AHRF) in Pediatrics
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to poor enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INOT-11
Record Dates: First submitted 2002-07-10; First posted 2002-07-11 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Respiratory Insufficiency; Anoxemia
Keywords: Acute hypoxemic respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia | interventions — Nitrogen; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Nitrogen gas
  Interventions: Drug: Nitrogen gas
- 1 (Experimental): Inhaled Nitric Oxide
  Interventions: Drug: inhaled nitric oxide

INTERVENTIONS:
Drug: Nitrogen gas — Nitrogen gas will be given at 5ppm until Day 28 or extubation
  Arms: 2
Drug: inhaled nitric oxide — inhaled nitric oxide will be given at 5 ppm until day 28 or extubation
  Other Names: INOmax®
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of nitric oxide for inhalation on the duration of mechanical ventilation in pediatric patients with AHRF.

DETAILED DESCRIPTION:
Patients will receive 5-ppm study gas (nitric oxide for inhalation or placebo) until Day 28 or extubation, whichever comes first. The following will be performed / recorded at specified times during the study: arterial blood gases, ventilator settings, methemoglobin, PRISM III score, and patient positioning. Selected centers will also be performing plasma cytokine assays, broncho-alveolar lavage fluid assays and a 6 month follow-up assessment.

ELIGIBILITY:
Inclusion criteria:

* Admitted to pediatric intensive care unit and have the diagnosis of acute respiratory failure
* 44 weeks post conceptional age to 16 years of age
* Oxygenation Index (OI) >=12 cm H2O/mmHg (as determined by two separate measurement taken 30 minutes to 4 hours apart)
* Recent chest x-ray (within 24 hours) showing at least unilateral infiltrations
* Mechanically ventilated <= 7 days

Exclusion criteria:

* Immunocompromised
* Received a bone marrow transplant
* Active oncological condition
* Persistent right to left intracardiac shunt
* Cardiovascular surgery within the last 14 days
* Status asthmaticus
* Decision by primary care physician not to provide full support
* Received treatment with nitric oxide for inhalation or other investigational medications within 24 hours prior to study initiation, participating in surfactant trials
* Chronically ventilated
* Pregnant

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
arterial blood gases | baseline through 24 hours and extubation

SECONDARY OUTCOMES:
methemoglobin | baseline, hour 4 and 24 hours
broncho-alveolar lavage fluid | baseline, 48 hours and day 5
Prone position | baseline then daily

CONTACTS AND LOCATIONS:
Overall Officials: James Baldassarre, MD, Study Director — Mallinckrodt
Locations (16):
- United States (16):
  - Chrildren's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Stanford, California
  - The Children's Hospital, Denver, Colorado
  - Nemours Children's Clinic, Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - University of Chicago, Children's Hospital, Chicago, Illinois
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - New York Presbyterian Hospital, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Pediatric Critical Care, Charlottesville, Virginia